CLINICAL TRIAL: NCT05626361
Title: Effect of Specialized Dysphagia Training on Knowledge and Competency of Nurses
Brief Title: Specialize Dysphagia Training and Knowledge/Competency of Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/13106 Raffa Mubeen
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Dysphagia
Keywords: Dysphagia; Swallowing disorder; Dysphagia screening; Nurses role; Assessment
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specialized Dysphagia training (Experimental): Power point presentation covering material related to nursing evaluation and caring of dysphagia patients. Stimulation session with nurses to practice screening skill
  Interventions: Other: Dysphagia training
- Reading material (Active Comparator): Reading material covering information related to nursing evaluation and caring of dysphagia patient
  Interventions: Other: Reading material

INTERVENTIONS:
Other: Dysphagia training — Training using PowerPoint and simulation. Training includes anatomy physiology, screening and management sections. Simulation will be used for practice. Reading material will also be provided
  Arms: Specialized Dysphagia training
Other: Reading material — Reading material provided to nurses covering knowledge related to nursing evaluation and caring for dysphagia patients
  Arms: Reading material

SUMMARY:
The aim of this research is to determine the effect of specialized dysphagia training on knowledge and competency of nurses.

ELIGIBILITY:
Inclusion Criteria:

* Nurses of both gender
* At least one year of experience
* Nurses working at Govt. hospital

Exclusion Criteria:

* Undergraduate nursed working as intern at hospital

Ages: 23 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Nurses Knowledge and competency regarding dysphagia scale | 1st day
  Change from base line, Nurses knowledge and competency regarding dysphagia scale is self developed scale. The scale include items related to anatomy physiology, risk factors, sign and symptoms, complications, screening, and management measured on 11 point scale.
Nurses Knowledge and competency regarding dysphagia scale | 3 months
  Change from base line to follow up of 3 months, Nurses knowledge and competency regarding dysphagia scale is self developed scale. The scale include items related to anatomy physiology, risk factors, sign and symptoms, complications, screening, and management measured on 11 point scale.

SECONDARY OUTCOMES:
The simulation Design scale | 1st day
  Changes from baseline, The simulation design scale is twenty item five point scale. It is used to evaluate design features of simulation. The instrument is divided into two parts: one part is about the presence of specific features in the simulation, while the other part is about the importance of those features to the learner. The rating of the specific features is from 1 to 5 where 1 is strongly disagree with the statement and 5 is strongly agree with the statement. Importance part is rated from 1 to 5 where 1 is not important and 5 is very important
Educational practice questionnaire | 1st day
  Changes from baseline, Educational practice questionnaire consists of sixteen items and is five point scale. It is used to measure educational practices. The rating of the educational practices is from 1 to 5 where 1 is strongly disagree with the statement and 5 is strongly agree with the statement. Importance part is rated from 1 to 5 where 1 is not important and 5 is very important
Student satisfaction and self confidence in learning | 1st day
  Changes from baseline, Student satisfaction and self confidence in learning is 13 item scale and is used to measure students satisfaction with simulation activity and self confidence in learning. Student satisfaction and self confidence in learning is rated from 1 to 5 where 1 is strongly disagree with the statement and 5 as strongly agree with the statement

CONTACTS AND LOCATIONS:
Overall Officials: Asghar Khan, PhD, Principal Investigator — Riphah International University; Raffa Mubeen, PhD*, Principal Investigator — Riphah International University
Locations (1):
- District Headquarters Hospital Chakwal, Chakwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No